CLINICAL TRIAL: NCT01794806
Title: Efficacy of Socket Grafting for Alveolar Ridge Preservation: A Randomized Controlled Trial
Brief Title: Efficacy of Socket Grafting for Alveolar Ridge Preservation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Osteogenics Biomedical (Industry)
Responsible Party: Principal Investigator, Gustavo Avila-Ortiz, Associate Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201301766
Record Dates: First submitted 2013-01-22; First posted 2013-02-20 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-07

CONDITIONS: Atrophy of Edentulous Alveolar Ridge
MeSH Terms: interventions — Tooth Extraction; Transplantation; Transplantation, Homologous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tooth extraction and grafting (Experimental): Tooth extraction and grafting with allograft
  Interventions: Procedure: Tooth extraction and grafting with allograft
- Tooth extraction (Sham Comparator): Tooth extraction
  Interventions: Procedure: Tooth extraction

INTERVENTIONS:
Procedure: Tooth extraction and grafting with allograft — Alveolar ridge preservation using a bone grafting material (allograft) and a synthetic dPTFE (dense Polytetrafluoroethylene) barrier membrane
  Other Names: Alveolar socket grafting
  Arms: Tooth extraction and grafting
Procedure: Tooth extraction — Minimally traumatic single-rooted tooth extraction
  Arms: Tooth extraction

SUMMARY:
The purpose of this study is to clinically and radiographically assess whether the use of a ridge preservation technique significantly minimizes alveolar ridge resorption following tooth extraction.

DETAILED DESCRIPTION:
Subjects requiring single-rooted tooth extractions and future tooth replacement therapy with implant-supported restorations will be recruited. Subjects will be randomly assigned to either a control (tooth extraction alone) or an experimental group (tooth extraction and ridge preservation using an allograft to fill the alveolar socket covered with a non-absorbable, dense polytetrafluoroethylene membrane [dPTFE]). Clinical linear measurements of the ridge (horizontal and vertical) will be obtained using a tooth-supported stent. Following extraction, primary closure of the socket will not be attempted. Subjects will be re-evaluated at 1 and 4 weeks. Implant placement surgery will be performed at 16 weeks. Clinical measurements will be repeated upon surgical re-entry. Cone beam computed tomographic (CBCT) scans will be obtained at baseline (after tooth extraction) and at 14 weeks (prior to implant placement) to assess alveolar ridge volumetric changes (primary outcome). Secondary outcome measures include changes in bucco-lingual and apico-coronal clinical measurements of the ridge and changes in modified wound healing index changes overtime. The influence of the thickness of the facial and lingual bone of the alveolar ridge and the width of the keratinized tissue on the remodeling of the ridge will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 75 years.
* Gender: No restriction.
* Subjects must require a single-rooted tooth extraction (Tooth deemed as periodontally and/or restoratively hopeless), except lower incisors and second premolars.
* Subjects must be able and willing to follow instructions related to the study procedures.
* Subjects must have read, understood and signed an informed consent form.

Exclusion Criteria:

* Reported allergy or hypersensitivity to any of the products to be used in the study.
* Severe hematologic disorders, such as hemophilia or leukemia.
* Active severe infectious diseases that may compromise normal healing.
* Liver or kidney dysfunction/failure.
* Currently under cancer treatment or within 18 months from completion of radio- or chemotherapy.
* Subjects who have a long-term history of oral bisphosphonate use (i.e. 10 years or more).
* Subjects with a history of IV bisphosphonates.
* Subjects with uncontrolled diabetes.
* Subjects with severe metabolic bone diseases, such as Paget's disease of bone, will be excluded.
* Pregnant women or nursing mothers.
* Smokers: Subjects who have smoked within 6 months of study onset.
* Concomitant medications: Subjects on concomitant drug therapy for systemic conditions that may affect the outcomes of the study will not be included in the study.

NOTE: Occasional, short-term use (7-14 days) of analgesics or common cold medications is permitted. Use of such medications will be reviewed and recorded by the investigator.

- Any other non-specified reason that from the point of views of the investigators will make a candidate not a suitable subject for the study (e.g. limited mouth opening).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2013-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Avila-Ortiz, DDS, MS, PhD, Principal Investigator — UI College of Dentistry
Locations (1):
- University of Iowa College of Dentistry - Craniofacial Clinical Research Center, Iowa City, Iowa, United States

REFERENCES:
- [Derived] Avila-Ortiz G, Gubler M, Romero-Bustillos M, Nicholas CL, Zimmerman MB, Barwacz CA. Efficacy of Alveolar Ridge Preservation: A Randomized Controlled Trial. J Dent Res. 2020 Apr;99(4):402-409. doi: 10.1177/0022034520905660. Epub 2020 Feb 12. PMID 32050833

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tooth Extraction and Grafting | Tooth Extraction
Started | 31 | 28
1 Week | 28 | 28
4 Weeks | 26 | 27
Completed | 26 | 27
Not Completed | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tooth Extraction and Grafting | Tooth Extraction | Total
Number analyzed (Participants) | 31 | 28 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 21 | 44
  >=65 years | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.46 (12.37) | 57.24 (11.82) | 57.84 (11.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 14 | 14 | 28
Region of Enrollment [Number; unit: participants]
  United States | 31 | 28 | 59

OUTCOME MEASURES:

1. Primary Outcome: Alveolar Ridge Volumetric Changes
Description: 3D reconstructions using radiographic data obtained at baseline and at 14 weeks after the intervention was utilized to calculate the reduction of bone volume that took place during the healing period in both groups
Time Frame: Baseline to Week 14 after tooth extraction
Measure: Mean (Standard Deviation); unit: percentage of volume change
Arm/Group | Tooth Extraction and Grafting | Tooth Extraction
Number analyzed (Participants) | 26 | 27
percentage of volume change | -8.36 (3.81) | -15.83 (4.48)

2. Secondary Outcome: Changes in Bucco-lingual Ridge Dimension
Description: Linear ridge width change at the bone crest
Time Frame: Baseline to Week 14 after tooth extraction
Measure: Mean (95% Confidence Interval); unit: millimeters
Arm/Group | Tooth Extraction and Grafting | Tooth Extraction
Number analyzed (Participants) | 26 | 27
millimeters | -1.0 [-1.49 to -0.64] | -1.8 [-2.10 to -1.26]

3. Secondary Outcome: Changes in Apico-coronal Ridge Dimension
Description: Linear ridge height change at the mid-facial aspect of the ridge
Time Frame: Week 14 after tooth extraction
Measure: Median (Inter-Quartile Range); unit: millimeters
Arm/Group | Tooth Extraction and Grafting | Tooth Extraction
Number analyzed (Participants) | 26 | 27
millimeters | -0.61 [-0.94 to -0.46] | -1.17 [-2.10 to -0.70]

ADVERSE EVENTS:
Arm/Group | Tooth Extraction and Grafting | Tooth Extraction
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/28
Other Adverse Events (participants affected / at risk) | 0/31 | 2/28
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tooth Extraction and Grafting (N=31) | Tooth Extraction (N=28)
Dry Alveolitis (Infections and infestations) | 0 (0) | 2 (2) — Dry Socket

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes